CLINICAL TRIAL: NCT04403945
Title: The Predictive Value of Sidestream Dark Field Imaging in Diabetic Nephropathy: a Observational Clinical Trial Evaluating the Predictive Value of SDF in DN
Brief Title: The Predictive Value of Sidestream Dark Field Imaging in Diabetic Nephropathy
Status: Completed | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Other Study IDs: PVSDFI-DN
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Microcirculation Detection in Diabetic Patients
Keywords: Type 2 Diabetes Mellitus; Sidestream dark field imaging; sublingual microcirculation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: healthy volunteers with normal fasting blood glucose and HbA1c, without hypertension, kidney diseases, or taking drugs that affects microcirculation
  Interventions: Device: Sidestream dark field(SDF) imagining
- Group 2: type 2 diabetic patients without microvascular complications like Diabetic nephropathy, diabetic retinopathy, diabetic foot or diabetic peripheral neuropathy
  Interventions: Device: Sidestream dark field(SDF) imagining
- Group 3: type 2 diabetic patients with diabetic nephropathy diagnosed by clinic or pathology.
  Interventions: Device: Sidestream dark field(SDF) imagining

INTERVENTIONS:
Device: Sidestream dark field(SDF) imagining — SDF imaging consists of a hand-held device that illuminates a region by surrounding a central light guide with concentrically placed light emitting diodes,which thus provide SDF illumination.

SUMMARY:
Diabetic microangiopathy refers to the pathological changes of arterioles, capillaries and venules in diabetic patients. Due to the impacts including glycol-metabolism disorder, disturbance of lipid metabolism, cytokine, oxidative stress and hemodynamic changes, the structure and function of microvessels are damaged accordingly. Diabetic nephropathy (DN) is one of the most common and serious chronic microvascular complications of diabetes, and becomes a leading cause of end-stage renal failure(ESRF). Presently, urinary albumin/creatinine ratio (UACR) is a widely accepted and relatively reliable indicator for early diagnosis of DN, however, there are 2/3 DN patients with normal albuminuria have decreased glomerular filtration rate (glomerular filtration rate, GFR) and abnormal structure of the kidney, one the other hand, the presence of albuminuria is associated with other vascular dysfunction and kidney disease other than DN, therefore its accuracy is increasingly being challenged.

Sidestream dark field(SDF) imagining technology, as an emerging way to visualize blood vessels, is evaluated in a semi-quantitative manner and provides an effective means to study structure and function of microcirculation. Different from biochemical markers like albuminuria, SDF provides a visual information about vessel structure, density, and quality of diffusion. At present the research of sublingual microcirculation by SDF technique is mainly applied to microcirculation monitoring in patients in the intensive care unit or laboratory animal models with acute hemorrhagic shock to assess the potential of being a tool of diagnosis and treatment prognostic indicator, no relevant research has been carried out to evaluate the predictive value of diabetic microangiopathy in literature so far.

Herein, the investigators designed the study based on SDF imaging to collect scientific data, thus providing strong support for the early assessment and diagnosis of diabetic nephropathy and possibly guiding individual therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

* age ranges from 18 to 70 years old
* signed informed consent

Exclusion Criteria:

* Younger than 18 years old or older than 70 years old
* Shock patients who have low blood pressure under 90/60mmHg
* Patients with mental abnormality who are uncooperative with this study
* Having difficulty in mouth opening
* Patients with Ketoacidosis
* Oral mucosal inflammation or injury, which could locally influence the sublingual microvasculature
* Pregnant or lactating women
* Refuse to sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We collected clinical data of 100 cases with T2DM who hospitalized in our treatment center from March 2019 to September 2020, and SDFI was taken properly.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
the comparison of the density of total length of the small perfusd vessels(PDV) in the acquisition window between the 3 groups | 21 months
  We use dark-field microcirculation microscopic observation System (Chinese Advanced Vessel Analyse Contrast System 4.0, C - AVA - C version 4.0) developed by Li Hua company to compare interesting parameters of vessels between the three groups. PVD is one of the parameters indicated of the perfused vessel density, calculated by the ratio of the length of small perfusion vessels to the visual field area (unit: mm/mm2)

SECONDARY OUTCOMES:
the comparison of The density of the total length of small vessels(TVD) in the area of the acquisition window between the 3 groups | 21 months
  We use dark-field microcirculation microscopic observation System (Chinese Advanced Vessel Analyse Contrast System 4.0, C - AVA - C version 4.0) developed by Li Hua company to compare interesting parameters of vessels between the three groups. TVD is one of the parameters indicated of the total vessel density, calculated by the ratio of the length of all small vessels to the visual field area (unit: mm/mm2)
the comparison of Proportion of De Backer density score between the 3 groups | 21 months
  The score is the result of counting the number of intersections of capillaries with predetermined grid lines and measurement of total capillary length relative to image surface are similarly reliable measures of functional capillary density
Correlation comparison: The correlation between SDF vascular parameters and the clinical data of the subjects was compared | 21 months
  Main clinical data:1. microalbuminuria；2.microalbuminuria creatinine ratio；3.Ankle brachial index；4.toe brachial index

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality, China